CLINICAL TRIAL: NCT05569499
Title: Evolution of Hematocrit in Burn Patients as a Marker of Fluid Management During Acute Phase
Brief Title: Hematocrit Evolution in Severe Burns
Acronym: HEREBUS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-13Obs-CHRMT
Record Dates: First submitted 2022-09-30; First posted 2022-10-06 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-09

CONDITIONS: Severe Skin Burns
MeSH Terms: conditions — Paresthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Burn-induced shock is described as being superimposed on sterile shock. with an increase in capillary permeability affecting healthy and burnt tissue and explains the formation of a large third sector.

Hematocrit is a criterion used historically to help adjust hydration in burn patients. This measurement due to its characteristics and accessibility suggests that it could be a good marker for monitoring hemodynamic resuscitation. The evolution of this parameter in relation to the conduct of volume resuscitation is assessed.

Thus, a retrospective, monocentric study is conducted at the Metz Burn Centre (France).

Inclusion criteria were admission to the intensive care unit of the Metz hospital between 01/04/2014 and 31/12/2021, for a Total Body Surface Area (TBSA) of at least 20%. The exclusion criteria were the presence of a burn involving a TBSA under 20%, minor patients, chemical, abrasion or radiation burns. Several clinical and paraclinical parameters have been reported and in particular the volumes of hydration and the variations in hematocrit during the first 24 hours. Measures of linear association between two continuous variables are calculated by the Pearson coefficient. The threshold of statistical significance was defined as a p-value of <0.05.

DETAILED DESCRIPTION:
Burn-induced shock is described as being superimposed on sterile shock. The inflammatory reaction secondary to tissue destruction leads to the release of multiple inflammatory mediators into the bloodstream, resulting in the development of systemic inflammatory response syndrome (SIRS). This is responsible for an increase in capillary permeability affecting healthy and burnt tissue and explains the formation of a large third sector.

The initial resuscitation of this state of shock differs from other management of shocked patients by the importance of its hypovolaemic side. Indeed, this is based on the evaluation of the filling needs through the Parkland formula defining the volume of hydration over twenty-four hours that should be administered. This guided and stereotyped haemodynamic resuscitation could lead to a state of fluid creep if it is not correctly monitored. Indeed, the importance of crystalloid solutions would lead to numerous complications such as pneumopathy or respiratory distress, cardiac failure or abdominal compartment syndrome. It is therefore necessary to adjust the fluid intake for the first twenty-four hours. This adjustment is made by means of various parameters including blood pressure and hourly diuresis. For some, the use of TEE, thermodilution or pulmonary artery catheterisation would allow more personalised and appropriate management.

Haematocrit is a criterion used historically to help adjust hydration in burn patients. Animal studies have shown it to be a good reflection of haemoconcentration caused by a burn. Haematocrit and haemoglobin levels change significantly downwards after a one litre saline filling in humans. The haematocrit has been shown to be a reliable reflection of hydration status in children and adults and can be used to assess the volume to be administered to correct dehydration states. Another criterion for monitoring haemodynamic resuscitation by haematocrit seems to be the availability of many biological tests in the initial phase of management of patients in shock. The measurement of haematocrit due to its characteristics and accessibility suggests that it could be a good marker for monitoring haemodynamic resuscitation in burn patients. The evolution of this parameter in relation to the conduct of volume resuscitation is assessed during the first twenty-four hours in severely burned patients.

A retrospective, monocentric study is conducted at the Metz Burn Centre (France). Various parameters were recorded: sex, age, weight (and its variations during the first 48 hours), height, TBSA, presence of cardiovascular comorbidities, IGS II, Baux Score, ABSI, BOBI, UBS score, origin of the burn, percentage of third degree, presence of inhalation, filling before admission and then hydration during the first 24 hours, the evolution of haematocrit, haemoglobin and albumin over the first 48 hours, hourly diuresis over the first 48 hours as well as the presence of mechanical ventilation (PAFI and its variations during the first 48 hours) or extra renal purification.

ELIGIBILITY:
Inclusion Criteria:

* Burns over 20% of Total Body Surface Area (TBSA)
* Hospitalization in Mercy Hospital (France) Intensive Care Unit

Exclusion Criteria:

* Age under 18 y
* chemical, abrasion or radiation burns

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: severly burned patients
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Hematocrit evolution | 24 hours following patient admission in intensive care unit
  Hematocrit level measured between the eighth and twenty-fourth hour minus the hematocrit level on admission

SECONDARY OUTCOMES:
Mortality in intensive care unit | at discharge of intensive care unit, average of 14 days
  mortality rate

CONTACTS AND LOCATIONS:
Overall Officials: Serge LE TACON, MD, Principal Investigator — CHR Metz Thionville Hopital de Mercy
Locations (1):
- CHR Metz-Thionville/Hopital de Mercy, Metz, France